CLINICAL TRIAL: NCT04827277
Title: A Prospective Randomized Clinical Trial Comparing Total Shoulder Arthroplasty vs Reverse Shoulder Arthroplasty in Patients >75 Years of Age
Brief Title: TSA Versus RSA in Patients >75
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JABB20D.949
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Total Shoulder Arthoplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Reverse total shoulder replacement (Active Comparator): Participants will receive a reverse total shoulder arthroplasty
  Interventions: Procedure: Reverse Total Shoulder Replacement
- Anatomic total shoulder replacement (Active Comparator): Participants will receive an anatomic total shoulder arthroplasty
  Interventions: Procedure: Anatomic Total Shoulder Replacement

INTERVENTIONS:
Procedure: Reverse Total Shoulder Replacement — Participants will be randomized to a reverse total shoulder replacement
  Arms: Reverse total shoulder replacement
Procedure: Anatomic Total Shoulder Replacement — Participants will be randomized to an anatomic total shoulder replacement
  Arms: Anatomic total shoulder replacement

SUMMARY:
Total shoulder arthroplasty (TSA) has proven to be a predictable and successful operation for the treatment of symptomatic glenohumeral osteoarthritis (GHOA) with an intact rotator cuff. Results after TSA have not been as good in cases with rotator cuff dysfunction, however. Early glenoid loosening, shoulder pain and the need for revision surgery has been all associated with rotator cuff deficiency. Even in cases without tears, fatty infiltration of the rotator cuff has been associated with inferior outcomes in TSA.

Advanced age has been shown to be associated with increased fatty infiltration of the rotator cuff in shoulders with primary osteoarthritis. Because of this, one may propose that surgeons should avoid the potential complications with TSA and perform RSA for patients with advanced age. It is thus the purpose of this study to evaluate the patient reported outcomes (PROs) of total shoulder arthroplasty (TSA) compared with reverse shoulder arthroplasty (RSA) in patients >75 years of age

ELIGIBILITY:
Inclusion Criteria:

* All patients (75 years of age) at the time of surgery
* Patient is willing to participate by complying with pre and postoperative visit requirements
* Patient is willing to consent for enrollment
* Patient has advanced imaging (CT or MRI) that demonstrates an intact rotator cuff

Exclusion Criteria:

* Patients under the age of 75
* Need for any structural graft for repair of the shoulder during surgery
* Current infection of the proximal humerus or scapula
* Proximal humerus fracture
* Inadequate or malformed bone that precludes adequate support for prosthesis (B2, B3, C Glenoid morphology)
* Neuromuscular disorder that does not allow control of the shoulder joint
* Significant injury to the brachial plexus
* Diagnosis of inflammatory arthropathy
* Preoperative diagnosis of full thickness rotator cuff tear
* >Goutallier Stage 1 rotator cuff atrophy
* Prior shoulder arthroplasty
* Non-functioning deltoid muscle
* Patients who are known drug or alcohol abuser, or have a psychological disorder as defined by the DSM4 that could affect follow-up care
* Patient is a prisoner
* Patients who are currently involved in any personal injury litigation, or worker's compensation claims.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative satisfaction | 2 years
  Investigators will be measuring whether there is an increase in participants satisfaction after surgery as assessed by the American Shoulder and Elbow Score (ASES)
Postoperative Satisfaction | 2 years
  Investigators will be measuring whether there is an increase in participants satisfaction after surgery as assessed by the Simple Shoulder Test (SST)
Postoperative Pain | 2 years
  Investigators will be measuring whether there is an increase in participants satisfaction after surgery as assessed by the Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States